CLINICAL TRIAL: NCT03674099
Title: Imatinib for Multiple Sclerosis (MS) Relapses - a Phase II, Randomised Study
Brief Title: Imatinib for Multiple Sclerosis (MS) Relapses
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tomas Olsson (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Sponsor-Investigator, Tomas Olsson, Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Imatinib MS
Record Dates: First submitted 2018-09-14; First posted 2018-09-17 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis relaps; Imatinib; Methylprednisolone
MeSH Terms: conditions — Multiple Sclerosis | interventions — Imatinib Mesylate; Methylprednisolone

STUDY DESIGN:
Intervention Model Description: Randomized, single-blinded, controlled.
Who Masked: Outcomes Assessor
Masking Description: Treating physician not blinded, evaluating physician blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imatinib (Experimental): Imatinib will be administered orally one tablet (400mg) twice daily, 800mg per day for 14 consecutive days.
  Interventions: Drug: Imatinib Mesylate
- Methylprednisolone (Active Comparator): Methylprednisolone will be administered once a day either in tablets; Medrol 1g per day or iv; Solumedrol 1000 mg per day, both for three consecutive days.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Imatinib Mesylate — Tablets 400 mg
  Arms: Imatinib
Drug: Methylprednisolone — 1 g tablets or infusion
  Arms: Methylprednisolone

SUMMARY:
To investigate if treatment with Imatinib results in a better outcome than standard care in form of Methylprednisolone(MP) after MS-associated relapses.

ELIGIBILITY:
Inclusion Criteria:

* An acute exacerbation, relapse, in persons with RRMS, either newly diagnosis or on treatment with one of the long-term immunomodulatory drugs, or possible MS where the diagnosis is supported by typical MRI or cerebrospinal fluid changes typical of MS (this enables inclusion of persons with a first neuroinflammatory bout, with high risk of developing MS before fulfilling the McDonald criteria for definite MS, or high risk for developing MS in the category clinically isolated syndrome (CIS)/possible MS with supporting MRI lesions and/or cerebrospinal fluid aberrations suggesting intra-thecal immunoglobulin synthesis with oligoclonal bands/and/or increased free Kappa Light chains. The relapse should be deemed to require relapse treatment by the investigator and affect a functional domain with a minimum of grade 2.
* 18-55 years of age
* Affection of any of the following EDSS sub-domains representing the targeted neurological deficit: 1. Visual function. grade 0-6, 2. Brain stem function grade 0-5. 3. Pyramidal function, grade 0-6. 4. Cerebellar function, grade 0-5. 5. Sensory function grade 0-6, and deterioration at least one step in any of these EDSS domains
* EDSS ≤ 6 before the acute exacerbation
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, if they are using effective methods of contraception during the study. Acceptable birth control methods are those with a failure rate of less than 1% per year when used consistently and correctly according to CTFG, September 2014 "Recommendations related to contraception and pregnancy testing in clinical trials". Such methods include:

  1. Combined (estrogen and progestogen containing hormonal contraception associated with inhibition of ovulation.

     * oral
     * intravaginal
     * transdermal
  2. progestogen-only hormonal contraception associated with inhibition of ovulation

     * oral
     * injectable
     * implantable
  3. intrauterine device (IUD)
  4. intrauterine hormone-releasing system (IUS)
  5. bilateral tubal occlusion
  6. total abstinence or vasectomized partner.

Exclusion Criteria:

* A pseudo-relapse should be excluded, as deemed by the experienced treating neurologist, and as evidenced by an active infection, likely with fever, with reappearing new signs and symptoms in a previously affected neurological function.
* Inability to provide informed consent
* Concomitant medication with drugs which may increase the plasma concentration of Imatinib - ketoconazole, itraconazole , erythromycin and clarithromycin
* Concomitant medication with drugs which may decrease the plasma concentration of Imatinib: dexamethasone, phenytoin, carbamazepin, rifampicin, phenobarbital, fosphenytoin, primidon, Hypericum perforatum (St John's wort).
* Female patients with childbearing potential, if pregnancy cannot be excluded by pregnancy test (urine point-of-care pregnancy test).
* Patient is participating in other interventional study
* General infection or any other condition judged by the treating neurologist to contra-indicate Imatinib
* Any laboratory deviation of general bodily functions such as kidney, or renal function judged to be of clinical significance by the treating neurologist constitutes an exclusion criteria.
* Patients with a positive Hepatitis B-DNA test result or serology indicating latent infection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Functional system score (FSS) change in the most worsened FSS after 28 days due to the acute relapse | 28 days
  The primary endpoint is mean change between baseline and day 28 in the most worsened FSS due to the acute relapse comparing MP and Imatinib. In case more than one domain is affected, priority of selected FSS should be in the following order: 1) Pyramidal, 2) Brain stem, 3) Cerebellar, 4) Visual, 5) Sensory. At least a two step deterioration due to neuroinflammatory bout should have occurred. Bowel and Cerebral domains will not be considered in the primary endpoints. The FSS is graded accordingly: 1. Visual function. Grade 0-6 2. Brain stem function grade 0-5 3. Pyramidal function, grade 0-6 4. Cerebellar function, grade 0-5 5. Sensory function grade 0-6 6. bowel/bladder function 7. Cerebral functions

SECONDARY OUTCOMES:
Functional system score (FSS) change between baseline and week 12 in the most worsened FSS due to the acute relapse | 12 weeks
  In case more than one domain is affected, priority of selected FSS should be in the following order: 1) Pyramidal, 2) Brain stem, 3) Cerebellar, 4) Visual, 5) Sensory. At least a two step deterioration due to neuroinflammatory bout should have occurred.
Mean expanded disability status scale (EDSS) change between baseline and day 28 | 28 days
  Calculation of EDSS summary score is based on the FSS score, from 0-5 with 0 representing normal neurological exam and 10 representing death by MS
Mean change in 9-hole peg test (evaluates upper limb function) between baseline and day 28 | 28 days
  Evaluates upper limb function
Mean change in timed 25- walk between baseline and day 28 | 28 days
Mean change in symbol digital modality test (SDMT) between baseline and day 28 | 28 days
  Evaluates cognitive function, with a score range of 0 to 110, with 110 representing the best cognitive function
Mean change in Multiple Sclerosis Impact Scale (MSIS-29; MS-specific quality of life (QoL) scale) between baseline and day 28 | 28 days
  The MISIS-29 consists of 29 items (composed of 20- item physical scale and a 9-item psychological scale), graded from 1-5 points with 5 indicating the most severe impact. The points for the two scales are individually summarized. The physical scale results in a sum with a range 20-100 , where 100 indicates the worse health. The psychological scale is similarly resulting in a range between to 9- 45, where 9 is the least and 45 is the worst.
Mean change in EQ5D (EuroQol 5 dimensions) (general QoL) between baseline and day 28. | 28 days
  EQ-5D is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression
Any difference in number of new brain MRI lesions at day 14 with regards to the baseline, comparing the two drugs | 14 days
Any difference in number of new brain MRI lesions at day 28 with regards to the baseline, comparing the two drugs | 28 days

CONTACTS AND LOCATIONS:
Locations (14):
- Rigshospitalet, Copenhagen, Denmark
- Germany (3):
  - Uniklinik Köln, Cologne
  - Hamburg-Eppendorf, Hamburg
  - UKSH Campus Kiel, Kiel
- Norway (4):
  - Haukeland sjukhus, Bergen
  - Akershus University Hospital, Lørenskog
  - Rikshospitalet, Oslo, Oslo
  - Ullevåls sjukhus, Oslo
- Sweden (6):
  - Karolinska Universityhospital, Huddinge, Huddinge, Stockholm County
  - Neurology Sahlgrenska Hospital, Gothenburg
  - Linköping University Hospital, Linköping
  - Akademiskt specialistcentrum, Stockholm
  - Karolinska Universitetssjukhuset, Solna, Stockholm
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No